CLINICAL TRIAL: NCT05435547
Title: Randomized Controlled Trial of Preoperative Corticosteroids in Autoimmune ThyroidDisease
Brief Title: Preoperative Corticosteroids in Autoimmune Thyroid Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Alexandria D. McDow, Assistant Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10009
Record Dates: First submitted 2022-01-25; First posted 2022-06-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Graves Disease; Hashimoto Disease
MeSH Terms: conditions — Graves Disease; Hashimoto Disease | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Steroids (Experimental): Will be given pre-operative corticosteroid regimen
  Interventions: Drug: Dexamethasone
- placebo (Placebo Comparator): Will be given Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Will take Dexamethasone pre-operatively
  Arms: Steroids
Drug: Placebo — Will take Placebo pre-operatively
  Arms: placebo

SUMMARY:
This study proposes to randomize patients about to undergo surgery for their autoimmune, inflammatory thyroid disease, and determine if a short course of corticosteroids decreases the inflammation of the gland and makes surgery less difficult.

ELIGIBILITY:
* Inclusion Criteria:

  ■ Graves' disease or Hashimoto's disease with positive thyroid autoantibodies (TgAb, TPO, TSI, and/or TRAb) undergoing total thyroidectomy for their disease.
* Exclusion Criteria:

  * Pediatric patients < 18
  * Prior treatment with RAI
  * Prior neck surgeries
  * Known diagnosis of thyroid cancer
  * Diabetic patients on medications
  * A history of adverse reactions to corticosteroids.
  * Patients on any immunosuppressive regimen (such as organ transplant patients or patients treated for other autoimmune conditions). This includes patients with recent history of steroid therapy, or a history of adverse reactions to corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Thyroid difficulty Scale score | Day of Surgery
  This scale is completed by the surgeon to assess the difficulty of a thyroid operation, and includes 4 parameters (vascularity, friability, mobility/fibrosis, and gland size). The scale ranges from 4 points (best outcome) - 20 points (worst outcome). Higher scores indicate a more difficult operation.

SECONDARY OUTCOMES:
Change in blood flow / vascularity | Pre-operative visit and Day of Surgery
  The surgeon will use ultrasound to assess the vascularity of the surgical area. Scoring is dependent on thyroid gland size, whether there is substernal extension, and the level of vascularity. The minimum score (2) indicates normal vascularity and normal gland size with no substernal extension. The maximum score (11) indicates extensive vascularity and large gland size with substernal extension.
Surgical complication of transient hypocalcemia | Two weeks post-operative and six weeks post-operative
  Number of subjects with transient hypocalcemia (calcium <8.5)
Surgical complication of permanent hypocalcemia | through study completion, or 6 months
  Number of subjects with permanent hypocalcemia (calcium <8.5)
Surgical complication of transient hypoparathyroidism | Two weeks post-operative and six weeks post-operative
  Number of subjects with Post-op PTH <10
Surgical complication of permanent hypoparathyroidism | through study completion, or 6 months
  Number of subjects with Post-op PTH <10
Surgical complication of recurrent laryngeal nerve palsy | Two weeks post-operative and six-weeks post-operative, if clinically indicated
  Vocal cord dysfunction will be evaluated through voice assessment and/or flexible laryngoscopy
Change in SF-20 at 6 weeks | Six weeks post-operative
  score ranges from 0 to 100, higher scores indicate better functioning or quality of life
Change in SF-20 at 6 months | through study completion, an average of 6 months
  score ranges from 0 to 100, higher scores indicate better functioning or quality of life
Tg | through study completion, an average of 6 months
  Tg, 1.3-31.8 ng/mL;
TgAB | through study completion, an average of 6 months
  TgAB, 0-4.0 IU/mL;
TPO | through study completion, an average of 6 months
  TPO AB 0-9.0 IU/mL;
TSI | through study completion, an average of 6 months
  TSI 0-0.54 IU/L;
TRAb | through study completion, an average of 6 months
  TRAb 0-1.75 IU/L
ThyPRO | through study completion, an average of 6 months
  0 points (best outcome) - 340 points (worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria McDow, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - IU Health North Hospital, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No